CLINICAL TRIAL: NCT06454409
Title: A Phase 1b Study of the Multi-Kinase Inhibitor Regorafenib in Combination With the BCL-2 Inhibitor Venetoclax Plus Azacitidine in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Regorafenib in Combination With Venetoclax and Azacitidine for the Treatment of Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: resources
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23713; NCI-2024-04611 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23713 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Myelodysplastic Syndrome/Acute Myeloid Leukemia; Recurrent Acute Myeloid Leukemia; Recurrent Myelodysplastic Syndrome; Refractory Acute Myeloid Leukemia; Refractory Myelodysplastic Syndrome
MeSH Terms: conditions — GATA2 Deficiency; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Azacitidine; Specimen Handling; regorafenib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (regorafenib, venetoclax, azacitidine) (Experimental): Patients receive regorafenib PO QD on days 1-21 of each cycle, venetoclax PO QD on days 1-21 of each cycle, and azacitidine IV over 10-40 minutes on days 1-7 of each cycle. Cycles repeat every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration during screening and on study as well as blood sample collection on study.
  Interventions: Drug: Azacitidine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: Regorafenib; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given IV
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Drug: Regorafenib — Given PO
  Other Names: BAY 73-4506; Regorafenib Anhydrous
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase Ib trial tests the safety, side effects, best dose and effectiveness of regorafenib in combination with venetoclax and azacitidine in treating patients with acute myeloid leukemia (AML) that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). Regorafenib is in a class of medications called kinase inhibitors. It works by blocking the action of an abnormal protein that signals cancer cells to multiply. This helps to slow or stop the spread of cancer cells. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking BCL-2, a protein needed for cancer cell survival. Azacitidine is in a class of medications called demethylation agents. It works by helping the bone marrow to produce normal blood cells and by killing abnormal cells. Giving regorafenib in combination with venetoclax and azacitidine may be safe, tolerable and/or effective in treating patients with relapsed or refractory AML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and tolerability of the multikinase inhibitor regorafenib in combination with the BCL2 inhibitor/BH3-mimetic venetoclax plus the hypomethylating agent azacitidine in patients with relapsed/refractory (R/R) acute myeloid leukemia (AML).

II. Determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of regorafenib when co- administered with venetoclax and azacitidine.

SECONDARY OBJECTIVES:

I. Evaluate the anti-leukemic activity, as assessed by overall response rate (ORR: complete remission [CR] + CR with incomplete hematologic recovery [CRi] + CR with partial hematologic recovery [CRh] + partial remission [PR]) within the first 28 days (cycle 1).

II. Evaluate the anti-leukemic activity, as assessed by complete remission (CR+CRi+CRh), overall response (ORR: CR+CRi+CRh+PR) and minimal residual disease (MRD)- rate and duration over the study period.

III. Estimate overall survival (OS), progression-free survival (PFS) and duration of response (DOR) rate at 6 months and 1 year.

EXPLORATORY OBJECTIVES:

I. Determine biomarkers that may be predictive of regorafenib activity in this combination.

II. To evaluate expression levels of VEGF, phosphatidylinositol-glycan (PIG), and soluble (s)VEGFR2 pre and post-treatment.

III. To evaluate changes in angiogenesis and inflammation pre and post treatment by gene expression.

IV. To characterize gene expression changes, including genes involved in the RAS/MAPK pathway, by ribonucleic acid (RNA) sequencing pre and post treatment with regorafenib when co-administered with venetoclax and azacitidine.

V. To evaluate changes in the gene mutation status of leukemic cells before and after treatment with regorafenib, azacitidine, and venetoclax.

VI. Evaluate changes to phosphorylated (phospho)-ERK after treatment with combination therapy.

OUTLINE: This is a dose-escalation study of regorafenib in combination with venetoclax and azacitidine followed by a dose-expansion study.

Patients receive regorafenib orally (PO) once daily (QD) on days 1-21 of each cycle, venetoclax PO QD on days 1-21 of each cycle, and azacitidine intravenously (IV) over 10-40 minutes on days 1-7 of each cycle. Cycles repeat every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration during screening and on study as well as blood sample collection on study.

After completion of study treatment, patients are followed up at 30 days then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Patients with histologically confirmed AML, according to World Health Organization (WHO) criteria, with refractory/relapsed (R/R) disease who are ineligible for therapies known to be effective for treatment of their AML

  * Patients with extramedullary disease may be included if they also have marrow involvement
  * Patients with acute promyelocytic leukemia (APL) will not be eligible
* Patients with R/R myelodysplastic syndrome (MDS)/AML, as defined by the presence of 10 - 19% blasts, are also eligible at the discretion of the principal investigator (PI)
* Fully recovered from the acute toxic effects (except alopecia) to ≤ grade 1 to prior anti-cancer therapy
* Ability to swallow pills
* White blood cells (WBC) ≤ 25 x 10^9/L prior to initiation of study therapy. Cytoreduction with hydroxyurea prior to treatment and/or during cycle 1 may be required (To be performed within 14 days prior to day 1 of protocol therapy)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (unless has Gilbert's disease) (To be performed within 14 days prior to day 1 of protocol therapy)
* Aspartate aminotransferase (AST) ≤ 3.0 x ULN (To be performed within 14 days prior to day 1 of protocol therapy)
* Alanine aminotransferase (ALT) ≤ 3.0 x ULN (To be performed within 14 days prior to day 1 of protocol therapy)
* Creatinine clearance of ≥ 45 mL/min per 24 hour urine test or the Cockcroft-Gault formula (To be performed within 14 days prior to day 1 of protocol therapy)
* International normalized ratio (INR) OR Prothrombin (PT) ≤ 1.5 x ULN (To be performed within 14 days prior to day 1 of protocol therapy)
* Activated partial thromboplastin Time (aPTT) ≤ 1.5 x ULN (To be performed within 14 days prior to day 1 of protocol therapy)
* Corrected QT interval by Fredericia (QTcF) ≤ 480 ms based on Fridericia's formula. (To be performed within 14 days prior to day 1 of protocol therapy) Note: To be performed within 28 days prior to day 1 of protocol therapy
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. (To be performed within 14 days prior to day 1 of protocol therapy)
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 4 months (males) and 7 months (females) after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Hematopoietic stem cell transplant within 100 days prior to day 1 of protocol therapy
* Chemotherapy, radiation therapy, biological therapy, immunotherapy within 14 days or five half-lives (whichever is shorter) prior to day 1 of protocol therapy with the following exceptions:

  * Subjects will be allowed to have been on venetoclax and/or azacitidine at screening and remain on it through treatment start
  * Hydroxyurea is allowed prior to treatment and through cycle 1 for control of rapidly progressing leukemia
* Strong and moderate CYP3A4 inducers and strong CYP3A inhibitors within 7 days prior to day 1 of protocol therapy
* Foods/supplements that are strong inhibitors or strong or moderate inducers of CYP3A (such as grapefruit, Seville oranges, starfruit and St. John's wort) within 3 days prior to initiation of and during study treatment
* Systemic steroid therapy > 10 mg/day (≤ 10mg/day prednisone equivalent ok) or any other form of immunosuppressive medication within 14 days. Inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent, are permitted. Steroids given for infusion prophylaxis or infusion reactions should not count towards this maximum
* Must not have received or planning to receive live vaccine while being on study or 4 weeks before and after completion of treatment
* Evidence or history of bleeding diathesis or coagulopathy
* Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) deep vein thrombosis or pulmonary embolism within 6 months of start of study treatment within 6 months of informed consent
* Presence of a non-healing wound, non-healing ulcer, or bone fracture
* Major surgical procedure or significant traumatic injury within 28 days before start of study medication
* Pleural effusion or ascites that causes respiratory compromise ( ≥ National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE] version 5.0 grade 2 dyspnea)
* Patients with blast phase chronic myeloid leukemia (CML)
* Patients with t(15;17) karyotypic abnormality or acute promyelocytic leukemia (French-American-British [FAB] class M3-AML)
* Active central nervous system (CNS) disease
* Active graft versus host disease (GVHD)
* Unstable cardiac disease as defined by one of the following:

  * Cardiac events such as myocardial infarction (MI) within the past 6 months
  * Uncontrolled atrial fibrillation or hypertension
* No measurable disease in the bone marrow
* Active diarrhea
* Gastrointestinal disorder that interferes with oral drug absorption such as malabsorption syndrome
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Uncontrolled active infection
* Clinically significant uncontrolled illness
* Diagnosis of Gilbert's disease
* Other active malignancy. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2030-09-06 (Estimated); Study Completion 2030-09-06 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to completion of cycle 1 (28 days)
  DLT will be defined as any toxicities classified as at least possibly related to the study treatment, that occur during cycle 1 and will be used for dose escalation/de-escalation/expansion decisions. Toxicity will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.
Incidence of adverse events (AEs) | Up to 30 days after last dose of study drug
  AEs will be graded according to the NCI CTCAE v 5.0 and reported by type, frequency, severity, attribution, time course, and duration.

SECONDARY OUTCOMES:
Complete remission (CR) rate | Up to 1 year
  Response will be determined using European LeukemiaNet criteria of Dohner et al. Response rates and Clopper-Pearson binomial confidence interval (CI) will be calculated for the CR (CR/ CR with incomplete hematologic recovery [CRi] / CR with partial hematologic recovery [CRh]) rate. CR rate will also be explored based on number/type of prior therapies.
Overall response rate (ORR) | Up to 1 year
  Response will be determined using European LeukemiaNet criteria of Dohner et al. Response rates and Clopper-Pearson binomial CI will be calculated for the ORR (CR/CRi/CRh/partial response [PR] / stable disease [SD]). ORR rate will also be explored based on number/type of prior therapies.
Minimal residual disease (MRD) | Up to 1 year
  MRD status will be determined by standard of care flow cytometry assay performed locally using a 0.01% blast threshold for positivity. MRD will be reported over the study period using both descriptive statistics and graphical methods.
Time to CR | At first dose of study drug to up to 1 year
  Time to CR will be defined as the time from first study dose to attainment of CR/ CRi/ CRh. Time to CR will be estimated using the product limit method of Kaplan-Meier.
Time to first response | At first dose of study drug to first documented response up to 1 year
  Time to first response will be defined as the time from first study dose to attainment of first documetned CR, CRi, CRh, morphologic leukemia-free state (MLFS) or PR. Time to first response will be estimated using the product limit method of Kaplan-Meier.
Duration of response (DOR) | At first response to relapse or death up to 1 year
  DOR will be defined as the time interval from the date of first documented response to the date of documented disease relapse or death whichever occurs first. DOR will be estimated using the product limit method of Kaplan-Meier.
Overall survival (OS) | At first dose of study drug to death up to 1 year
  OS will be defined as the time interval from the date of first study dose to the date of death from any cause. OS will be estimated using the product limit method of Kaplan-Meier.
Progression-free survival (PFS) | At first dose of study drug to relapse, progression, or death up to 1 year
  PFS will be defined as the time interval from the date of first study dose to the date of first documented disease relapse/progression or death from any cause, whichever occurs first. PFS will be estimated using the product limit method of Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Koller, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States